CLINICAL TRIAL: NCT00112268
Title: Quitlink : A Leveraging Solution to Tobacco Counseling
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Virginia Ambulatory Care Outcomes Research Network (Other)
Organization: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: 1R21HS014854-01 (AHRQ); 1R21HS014854-01 (AHRQ)
Record Dates: First submitted 2005-06-01; First posted 2005-06-02 (Estimated); Last update posted 2006-10-27 (Estimated); Status verified 2006-10

CONDITIONS: Smoking
Keywords: randomized controlled trial; primary health care; smoking cessation
MeSH Terms: conditions — Smoking; Smoking Cessation

INTERVENTIONS:
Behavioral: QuitLink (office support system for quit line referral)

SUMMARY:
Primary: To test whether the delivery of A3-5 smoking cessation counseling (Assess, Assist, Arrange) in primary care offices is enhanced by a system that couples (1) an expanded vital sign intervention with (2) fax referral of preparation-stage patients for telephone counseling and (3) feedback to the provider. The question will be examined in a randomized trial, with practices as the unit of analysis and with a control intervention consisting of a conventional vital sign intervention. The experiment will therefore compare what intervention and control practices accomplish beyond simply identifying patients who use tobacco.

Secondary: To assess contextual factors that might affect implementation of the intervention and account for its ultimate success or failure. In particular, to assess: (1) environmental and practice-level factors that affect practices' ability to successfully implement and use the intervention and; (2) patient characteristics beyond readiness to change (i.e., age, gender, race/ethnicity) that affect willingness to use the quit line and complete counseling.

DETAILED DESCRIPTION:
Among the most important evidence-based interventions in primary care is to offer counseling and pharmacotherapy to patients who use tobacco, but studies suggest that only a fraction of tobacco users receive this assistance. Office systems and other strategies can improve counseling rates but are not widely adoptable in primary care. We propose a novel solution that couples a simple office system, which is widely adoptable, with a form of third-party counseling (telephone quit lines) that most practices can access in the United States. Specifically, the three-part intervention includes (1) an in-office expanded "vital signs" intervention that prompts nurses (or medical assistants) to determine tobacco use status, offer brief advice, and assess readiness to quit as vital signs are obtained; (2) inviting preparation-stage tobacco users to obtain proactive telephone counseling (provided by the American Cancer Society) comprising three 30-minute sessions scheduled at the patient's convenience; and (3) feedback from the Society to the practice, including fax requisitions for prescription aids for quit attempts, progress reports on the results of counseling, and quarterly aggregate analyses of practice and clinician team referral outcomes. The Virginia Ambulatory Care Outcomes Research Network will partner with the American Cancer Society to test this strategy in a randomized controlled trial conducted at 16 primary care practices in Virginia. Because existing dissemination strategies serve mainly to increase identification of tobacco users and sometimes to increase brief advice, our primary outcome measure will be the proportion of tobacco users who receive substantive assistance: Assess, Assist, and Arrange of the 5As. Given the widening availability of state and national quit line programs, our model for referrals and bidirectional communication with primary care could markedly augment the effectiveness of both primary care and quit lines in promoting tobacco cessation and provide an attractive alternative for clinicians who lack the time and resources to provide effective counseling.

ELIGIBILITY:
Inclusion Criteria:

* Current use of tobacco
* Age 18 or older
* Visit with a clinician that day
* Patient at one of the 16 practices in the study

Exclusion Criteria:

* Unable to participate in a self-administered exit survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3200
Dates: Start 2005-06; Study Completion 2006-07

PRIMARY OUTCOMES:
Whether the intervention increases the proportion of tobacco users (age 18 and older) who receive help within the domains of A3-5 (Assess, Assist, and/or Arrange) at the index office visit, as reported by exiting patients

SECONDARY OUTCOMES:
The frequency with which tobacco users are identified (Ask) and advised to quit (Advise)
The proportion of patients in the preparation stage who consent to telephone counseling
How recipients of A1-2, A3-5, and the offer of telephone counseling differ by age, gender, doctor seen, and reason for visit
The proportion of consenting patients who are contacted by American Cancer Society (ACS) counselors within 2 weeks of referral
The proportion who completed three counseling sessions

CONTACTS AND LOCATIONS:
Locations (1):
- Virginia Ambulatory Care Outcomes Network (ACORN), Richmond, Virginia, United States

REFERENCES:
- [Derived] Rothemich SF, Woolf SH, Johnson RE, Devers KJ, Flores SK, Villars P, Rabius V, McAfee T. Promoting primary care smoking-cessation support with quitlines: the QuitLink Randomized Controlled Trial. Am J Prev Med. 2010 Apr;38(4):367-74. doi: 10.1016/j.amepre.2010.01.008. PMID 20307804